CLINICAL TRIAL: NCT00916695
Title: Everolimus-Eluting Stent in the Treatment of Bifurcation Lesions: Comparison of Main Vessel Stent to Main Vessel and Side Branch Stent
Brief Title: Everolimus-Eluting Stent for Bifurcation Coronary Lesions: Comparison of Simple Versus Complex Techniques
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Fernando Martín Burrieza, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XV02RS; XV02RS
Record Dates: First submitted 2009-06-01; First posted 2009-06-09 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Coronary Artery Disease
Keywords: Stents; Angioplasty; Coronary Artery Disease; Bifurcation Coronary Lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complex PCI strategy for bifurcation coronary lesions (Active Comparator): Stenting main vessel and T-stenting for the side branch
  Interventions: Device: Xience V Everolimus Eluting Coronary Stent System. Abbott Laboratories. Abbott Park, Illinois, U.S.A.
- Simple PCI strategies for bifurcation coronary lesions (Active Comparator): Stenting main vessel, with provisional stenting for the side branch.
  Interventions: Device: Xience V Everolimus Eluting Coronary Stent System. Abbott Laboratories. Abbott Park, Illinois, U.S.A.

INTERVENTIONS:
Device: Xience V Everolimus Eluting Coronary Stent System. Abbott Laboratories. Abbott Park, Illinois, U.S.A. — Complex PCI strategy for bifurcation: After optional pre-dilation of one or both vessels (main and side branch), and subsequent implanting of the stent in the main vessel, the side branch is approached by implanting a new stent as T technique.
  Simple PCI strategy for bifurcation: After optional pre-dilation of one or both vessels (main and side branch), a stent is deployed at main vessel. Side branch is approached by using provisional T stenting technique.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the treatment of true bifurcation lesions with the XIENCE V stent using the simple strategy (stent in main vessel and provisional T-stenting in the side branch) compared to the complex strategy (stent in main vessel and T-stenting in the side branch).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* True Bifurcation lesion (Medina classification 1-1-1), in at least one main coronary vessel. Diameter of main vessel between 2,5-4mm, and diameter of side branch 2mm or greater.

Exclusion Criteria:

* Significant left main stenosis.
* ST elevation myocardial infarction < 48 h.
* Thrombus burden target lesion.
* Ejection Fraction < 30%.
* Severe Renal Insufficiency (creatinine > 3 mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rate of binary angiographic restenosis (in main vessel and side branch) in the simple versus complex strategy groups | 9 months

SECONDARY OUTCOMES:
Combined rate of events (cardiac death, myocardial infarction and TLR) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Federico Gimeno, MD, Principal Investigator — Hospital Clinico Universitario Valladolid; Bruno Garcia, MD, Principal Investigator — Hospital Valle de Hebron. Barcelona; Ramiro Trillo, MD, Principal Investigator — Hospital Clínico Santiago; Jose Moreu, MD, Principal Investigator — Hospital Virgen de la Salud; Javier Goicolea, MD, Principal Investigator — Hospital Puerta de Hierro, Madrid; Raul Moreno, MD, Principal Investigator — Hospital Universitario La Paz; Jose F Diaz, MD, Principal Investigator — Hospital Juan Ramon Jimenez. Huelva; Jose M Hernandez, MD, Principal Investigator — Hospital Clinico de Malaga; Ramon Lopez-Palop, MD, Principal Investigator — Hospital San Juan. Alicante; Mariano Valdes, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca; Pascual Bordes, MD, Principal Investigator — Hospital Universitario. Alicante; Jose R Rumoroso, MD, Principal Investigator — Hospital Galdakao. Vizcaya
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - University Hospital Virgen Macarena, Seville, Seville